CLINICAL TRIAL: NCT07091188
Title: A Culturally Adapted Digital Intervention to Promote Maternal Care Utilization Using Multifaceted Approaches (CALCIUM) Among an Ethnic Minority Community in China
Brief Title: A Culturally Adapted Digital Intervention to Promote Maternal Care Utilization Using Multifaceted Approaches
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiayao Xu (Other)
Responsible Party: Sponsor-Investigator, Jiayao Xu, Postdoctoral Researcher, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ZGL202408-7
Record Dates: First submitted 2025-07-06; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Antenatal Care; Pregnancy Complications; Pregnancy Outcomes
Keywords: antenatal care; ethnic minority; digital health; health education
MeSH Terms: conditions — Pregnancy Complications; Health Education | interventions — Capacity Building

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Interventions including digital health education via social media platform, capacity building for healthcare providers and economic incentives for village doctors will be applied
  Interventions: Behavioral: Health education, capacity building and economic incentives
- Control group (No Intervention): No intervention will be applied

INTERVENTIONS:
Behavioral: Health education, capacity building and economic incentives — 1. Social media platform-based for health education. Pregnant women in the same gestational month will be invited to join specific WeChat group chats tailored to their similar health education and management needs.
  2. Capacity building. ANC providers at township hospitals will participate in short-term, small-class training courses designed to cover essential aspects of antenatal care prior to the intervention with the pregnant women.
  3. Economic incentives. To encourage ANC attendance, a monetary reward system will be implemented for village doctors every time they successfully identify and invite a newly pregnant woman to initiate her ANC visit.
  Arms: Intervention group

SUMMARY:
Maternal healthcare utilization is crucial for reducing maternal mortality, yet remains low in many underserved regions. The CALCIUM intervention, a culturally tailored, digital platform-integrated intervention, was developed to promote antenatal care (ANC) and institutional deliveries in Liangshan Yi Autonomous Prefecture, an ethnic minority community in China. The CALCIUM intervention was developed to address barriers including limited healthcare awareness, traditional norms and low-quality services. This intervention will evaluate the effectiveness, and cost-effectiveness of improving maternal healthcare utilization and pregnancy outcomes in an ethnic minority community.

DETAILED DESCRIPTION:
A cluster quasi-randomised control trial will be conducted in two counties, Xide and Yuexi, in Liangshan Yi Autonomous Prefecture, Sichuan province, China. In total, 12 towns will be randomly selected from each of the two counties (i.e., Yuexi and Xide). Within each county, the selected towns will be randomly and evenly assigned to the intervention and control groups. In each town, 80 newly pregnant women will be invited to participate. The comprehensive intervention was designed based on the Behaviour Change Wheel (BCW) including digital health education via social media platform, capacity building for healthcare providers and economic incentives for village doctors. Primary outcomes include the rates of hospital delivery and ANC utilization. Secondary outcomes include participants' pregnancy-related diseases and pregnancy outcomes. Primary and secondary outcomes will be collected through the local maternal and newborn health monitoring system. Sociodemographic and process information will be gathered through postpartum interviews. A logistic mixed model with an intention-to-treat approach will be used to evaluate the effectiveness of the intervention. Additionally, intervention costs and cost-effectiveness will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women

Exclusion Criteria:

* Not pregnant women

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1920 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Rates of Hospital Deliveries and Completion of Five Antenatal Care Visits | Data will be collected at the end of the pregnancy
  The primary outcome includes the rate of maternal care utilization, including the rate of hospital delivery and ANC utilization. According to the National Basic Public Health Service Specifications, pregnant women are advised to have their first ANC visit by the 13th week of gestation, with subsequent visits recommended during the 16-20, 21-24, 28-36, and 37-40 week periods. Timely initiation of ANC is defined as pregnant women completing their first ANC visit by the 13th week of gestation. Timely completion of five ANC visits is defined as pregnant women completing all five recommended ANC visits within the specified timeline. ANC utilization is measured by the completion of five ANC visits, the timely completion of five ANC visits, and timely initiation of ANC. The maternal and newborn health monitoring system collects routine information related to ANC utilization, place of delivery, maternal outcomes, and birth outcomes. Data will be sourced from this system.

SECONDARY OUTCOMES:
Rate of Negative Pregnancy Outcomes | Data will be collected at the end of the pregnancy
  Participants' negative pregnancy outcomes, such as maternal death, neonatal death, postpartum haemorrhage, perinatal asphyxia, preterm birth (PTB), large for gestational age (LGA), small-for-gestational age (SGA), congenital malformations and neonatal intensive care unit admission.
Rate of Pregnancy-Related Diseases | Data will be collected from pregnancy through the end of the study, with an average follow-up duration of one year
  Pregnancy-related disorders, such as gestational anaemia, gestational hypertension, preeclampsia and gestational hyperglycaemia will be recorded.
Number of Tests Conducted | Data will be collected from pregnancy through the end of the study, with an average follow-up duration of one year
  The number of tests conducted for full blood count, blood pressure measurement, Down Syndrome screening, Nuchal Translucency screening, and 3D/4D ultrasound during ANC will be collected.

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to privacy considerations and data minimization principles.